CLINICAL TRIAL: NCT04699682
Title: Carriage Clearance of Emerging Highly Resistant Bacteria in Chronic Dialysis Patients
Acronym: DIACOBHR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DIACOBHR
Record Dates: First submitted 2020-12-30; First posted 2021-01-07 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Chronic Kidney Diseases; Dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): During follow-up visits, as part of this research, additional stool samples are taken every month (M1 to M12).
  Interventions: Other: Control
- BHR Case (Experimental): During follow-up visits, compared to the usual management of patients with BHRe (monthly sampling for 6 consecutive months), additional samples are taken as described below:
  - stool samples taken at different times:
  * every 7 days during the first month (M1)
  * every 14 days for the following months until the end of the patient's participation (M2 to M12).
  Interventions: Other: BHR Case

INTERVENTIONS:
Other: Control — During follow-up visits, as part of this research, additional stool samples are taken every month (M1 to M12).
  Arms: Control
Other: BHR Case — During follow-up visits, compared to the usual management of patients with BHRe (monthly sampling for 6 consecutive months), additional samples are taken as described below:
  - stool samples taken at different times:
  * every 7 days during the first month (M1)
  * every 14 days for the following months until the end of the patient's participation (M2 to M12).
  Arms: BHR Case

SUMMARY:
The propias, and more recently the update of the recommendations relating to the control of the spread of bacteria highly resistant to emerging antibiotics issued by the High Council of Public Health (December 2019), recommend the implementation of measures to maintain the rate of Carbapenemase-producing Enterobacteriaceae (EPC) such as Klebsiella pneumoniae (K. pneumoniae) isolated from bacteremia in healthcare establishments in France at less than 1%, and that of Vancomycin Resistant Enterococcus (VRE) belonging to Enterococci Resistant to Glycopeptides (ERG) such as Enterococcus faecium isolated from bacteremia in health establishments in France at less than 1% also. At the same time, the prevalence of colonized patients is increasing. One of the recommended measures concerns the fight against cross transmission.

Due to the high technicality of the treatments, the risks of cross-transmission are very high and present at each stage of the dialysis procedure. Screening and isolation of patients colonized with emerging Highly Resistant Bacteria (BHRe) is essential to avoid their spread and the risk of infection with these germs.

Screening is done using rectal swabs. If the patient is found to be a carrier of BHRe, he should be isolated. Isolation is made more difficult in the hemodialysis room due to their architectural configuration, the organization of care and the chronicity of the patients. Patients have a monthly sample.

The isolation is allowed after obtaining six consecutive negative rectal swabs, the number of which has been arbitrarily defined. Indeed, the negativation of the samples does not confirm the disappearance of the carriage (that is to say the presence of BHRe), hence the need to repeat them. Persistence of colonization at a rate below the detection limit is possible. With for corollaries:

* Isolation which could be lifted more quickly in the event of real disappearance of the strain since the investigators know that a prolonged period of isolation can lead to a loss of opportunity for the patient and the investigators know its impact for the patient, on the operation of the service and its cost, with in particular the increase in withdrawals.
* Isolation lifted too early in the event of persistent carriage with risk of secondary transmission.

The interest of this study is to determine the clearance of the carriage of BHRe, i.e. their disappearance, in the chronic dialysis patient and to define, secondly, the factors associated with the prolonged carriage corresponding to the presence of bacteria for more than 3 months. , and elements of answer concerning the early disappearance of the EPC in the event of co-colonization by ERG and EPC. The follow-up of this carriage for 1 year will make it possible to evaluate the relapse corresponding to the reappearance of the bacteria previously identified, the recolonization corresponding to the acquisition of a new BHR, or the reinfection corresponding to an infection with a new highly resistant bacterium.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years old)
* Patient with stage V chronic renal failure, treated by chronic dialysis (hemodialysis or peritoneal dialysis) and monitored at AURA Paris (AURA Paris Plaisance Dialyse and hospitalization, AURA Nord, AURA Corentin Celton, AURA Bichat)
* Patient affiliated to a health insurance plan
* French-speaking patient
* Patient who has given free, informed and written consent

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under legal protection
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2024-01-14 (Estimated); Study Completion 2025-03-14 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with disappearance of Carriage of bacteria | Year 1
  This outcome corresponds to the disappearance of the carriage of the emerging highly resistant bacteria over the follow-up period of one year.

SECONDARY OUTCOMES:
Prevalence of BHR carriage | Year 1
  This outcome corresponds to the proportion of patients with emerging highly resistant bacteria.
Comparison of Prevalence of BHR carriage between the 2 groups | Year 1
  This outcome corresponds to the comparison of carriage of emerging highly resistant bacteria between case patients and control patients.

CONTACTS AND LOCATIONS:
Overall Officials: Cecile BOURGAIN, MD, Principal Investigator — AURA Paris Plaisance
Locations (5):
- France (5):
  - AURA Corentin Celton, Paris, Groupe Hospitalier Paris Saint-Joseph
  - AURA Paris Plaisance, Paris, Groupe Hospitalier Paris Saint-Joseph
  - AURA Paris Site de Saint Ouen, Paris, Groupe Hospitalier Paris Saint-Joseph
  - Groupe Hospitalier Paris Saint-Joseph, Paris, Groupe Hospitalier Paris Saint-Joseph
  - AURA Bichat, Paris, Groupe Hospitalier Paris Saint-Joseph

REFERENCES:
- [Result] Fournier S, Brossier F, Fortineau N, Gillaizeau F, Akpabie A, Aubry A, Barbut F, Chedhomme FX, Kassis-Chikhani N, Lucet JC, Robert J, Seytre D, Simon I, Vanjak D, Zahar JR, Brun-Buisson C, Jarlier V. Long-term control of vancomycin-resistant Enterococcus faecium at the scale of a large multihospital institution: a seven-year experience. Euro Surveill. 2012 Jul 26;17(30):20229. PMID 22856512
- [Result] Davido B, Moussiegt A, Dinh A, Bouchand F, Matt M, Senard O, Deconinck L, Espinasse F, Lawrence C, Fortineau N, Saleh-Mghir A, Caballero S, Escaut L, Salomon J. Germs of thrones - spontaneous decolonization of Carbapenem-Resistant Enterobacteriaceae (CRE) and Vancomycin-Resistant Enterococci (VRE) in Western Europe: is this myth or reality? Antimicrob Resist Infect Control. 2018 Aug 13;7:100. doi: 10.1186/s13756-018-0390-5. eCollection 2018. PMID 30123500
- [Result] Zahar JR, Garrouste-Orgeas M, Vesin A, Schwebel C, Bonadona A, Philippart F, Ara-Somohano C, Misset B, Timsit JF. Impact of contact isolation for multidrug-resistant organisms on the occurrence of medical errors and adverse events. Intensive Care Med. 2013 Dec;39(12):2153-60. doi: 10.1007/s00134-013-3071-0. Epub 2013 Aug 31. PMID 23995982